CLINICAL TRIAL: NCT01142401
Title: A Randomized Phase II Study of Fulvestrant vs. Fulvestrant in Combination With Bortezomib in Women With ER Positive Metastatic Breast Cancer
Brief Title: Fulvestrant With or Without Bortezomib in Patients With Inoperable Locally Advanced or Metastatic Estrogen Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-03000; NCI-2012-03000 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000674542; 10-01555; AECM-000248; 10-03-055; 8457 (Other: Montefiore Medical Center - Moses Campus); 8457 (Other: CTEP); N01CM00070 (NIH); N01CM00099 (NIH); N01CM62204 (NIH); N01CM62207 (NIH); P30CA013330 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Breast Carcinoma; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Bortezomib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (fulvestrant) (Experimental): Patients receive fulvestrant IM on day 1 (days -14, 1, and 15 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may crossover to arm C.
  Interventions: Drug: Fulvestrant; Other: Laboratory Biomarker Analysis
- Arm B (fulvestrant, bortezomib) (Experimental): Patients receive fulvestrant as in arm A and bortezomib IV on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Fulvestrant; Other: Laboratory Biomarker Analysis
- Arm C (fulvestrant, bortezomib) (Experimental): Patients receive fulvestrant IV on day 1 and bortezomib IM on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Fulvestrant; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
  Arms: Arm B (fulvestrant, bortezomib); Arm C (fulvestrant, bortezomib)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well fulvestrant works with or without bortezomib in treating patients with estrogen receptor positive breast cancer that has spread to other places in the body and cannot be removed by surgery. Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by lowering the amount of estrogen the body makes. Bortezomib may stop the growth of breast cancer cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. It is not yet known whether fulvestrant is more effective with or without bortezomib in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the addition of bortezomib to fulvestrant improves median progression free survival (PFS) compared with fulvestrant alone in postmenopausal women with estrogen receptor (ER)-positive locally advanced inoperable or metastatic breast cancer who have disease that is resistant to aromatase inhibitor therapy (Arms A versus [vs.] B).

SECONDARY OBJECTIVES:

I. To determine if the addition of bortezomib to fulvestrant improves the clinical benefit rate (defined as objective response plus stable disease for at least 24 weeks from day +1).

II. To determine the percent of patients, treated with fulvestrant alone and fulvestrant plus bortezomib, who remain progression-free 24 weeks from day +1 (Arms A vs. B).

III. To determine the overall survival of patients treated with fulvestrant alone and fulvestrant plus bortezomib (Arms A, B, C).

IV. To determine the adverse event profile in patients treated with fulvestrant alone and fulvestrant plus bortezomib (Arms A, B, C).

V. To determine the clinical benefit rate at 12 and 24 weeks of fulvestrant plus bortezomib in patients who have progressed on the fulvestrant alone arm and crossover to receive the combination (Arm C).

TERTIARY OBJECTIVES:

I. To perform an exploratory analysis of the effects of bortezomib (plus fulvestrant) in intratumoral nuclear/cytoplasmic ER ratio, unfolded protein response (BiP), apoptosis (cleaved caspase 3), B-cell chronic lymphocytic leukemia (CLL)/lymphoma 2 (Bcl-2) phospho c-Jun N-terminal kinase (JNK) in patients with tumors accessible to biopsy who consent to optional post-treatment biopsy.

II. To determine with cyclin D1 expression in pretreatment tumor specimens (from metastatic disease or the primary tumor if the former is not available) is predictive of clinical benefit with fulvestrant-bortezomib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms (Arms A or B).

ARM A: Patients receive fulvestrant intramuscularly (IM) on day 1 (days -14, 1, and 15 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may crossover to arm C.

ARM B: Patients receive fulvestrant as in arm A and bortezomib intravenously (IV) on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive fulvestrant IM on day 1 and bortezomib IV on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY CRITERIA FOR ARM A AND ARM B
* Patients must have histologically or cytologically confirmed ER+ positive breast cancer
* Patients must be postmenopausal, defined as: (1) a history of at least 12 months without spontaneous menstrual bleeding, (2) prior bilateral salpingo-oophorectomy, with or without hysterectomy, (3) age >= 55 years with a prior hysterectomy with or without oophorectomy, (4) age < 55 years with a prior hysterectomy without oophorectomy or unknown status, with a documented follicle-stimulating hormone (FSH) level in postmenopausal range within 4 week s of registration, (5) receiving a gonadotropin releasing hormone analog (GnRH) to suppress ovarian function (eg, goserelin 3.6 mg every [q] 4 weeks)
* Patients must have stage IV disease or inoperable locally advanced disease
* Patients may have measurable disease only, non-measurable disease only, or both (Response Evaluation Criteria in Solid Tumors [RECIST 1.1]); it is anticipated that at least 50% of patients will have only non-measurable disease
* Patients are required to have disease that is resistant to aromatase inhibitor (AI), which is defined either as relapse while receiving adjuvant A.I. therapy (ie, anastrazole, letrozole, or exemestane), and/or disease progression after one or more A.I.s for metastatic disease; prior exposure to more than one AI is permitted
* Patient may have had prior tamoxifen but are not required to
* Patients may have received up to one prior chemotherapy regimen for metastatic disease
* Patients may have received prior bevacizumab
* Patients who have received up to 2 doses of fulvestrant given within a 4 week period prior to registration are eligible; the interval between the first fulvestrant dose and registration must be 6 weeks or less; patients may have received EITHER 250 mg or 500 mg of fulvestrant previously; if the patient has received 250 mg, they will receive the 500 mg loading dose on study day -14; if they already received 500 mg, they will begin the study on day +1
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must be disease-free of prior invasive malignancies for >= 5 years with the exception of: curatively-treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* ELIGIBILITY CRITERIA FOR ARM C
* Previously met all eligibility criteria for arms A and B and registered on trial to arm A (fulvestrant alone)
* Disease progression on arm A and agreeable to crossover to arm C
* Has received no intervening therapy (ie, alternative endocrine therapy, chemotherapy, biologic therapy) between disease progression on arm A and registration an arm C
* ECOG performance status 0-2
* Tumor measurements (eg, computed tomography [CT] scan of chest/abdomen/pelvis) within 4 weeks of registration to arm C
* Leukocytes >= 3,000/mcL, within 2 weeks of registration on arm C
* Absolute neutrophil count >= 1,500/mcL, within 2 weeks of registration on arm C
* Platelets >= 100,000/mcL, within 2 weeks of registration on arm C
* Total bilirubin within normal institutional limits, within 2 weeks of registration on arm C
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal, within 2 weeks of registration on arm C
* Creatinine within normal institutional limits, within 2 weeks of registration on arm C OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal, within 2 weeks of registration on arm C

Exclusion Criteria:

* EXCLUSION CRITERIA FOR ARM A AND ARM B
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* Presence of rapidly progressive, life-threatening metastases; this includes patients with extensive hepatic involvement (> 50% of the liver involved), symptomatic lymphangitic metastases, or brain or leptomeningeal involvement
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib or fulvestrant
* Patients who are concomitantly receiving bortezomib and drugs that are inhibitors or inducers of cytochrome P450 3A4 should be closely monitored for either toxicities or reduced efficacy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who have previously received fulvestrant
* Patients who have previously received bortezomib
* Concomitant anticancer treatment with the following exceptions: (1) bisphosphonates for bone metastases, (2) a GnRH analog is permitted if the patient had progressive disease on a GnRH analog plus a selective estrogen receptor modulators (SERMs) or an AI; the GnRH analog may continue but the SERM or AI must be discontinued
* Grade 2 or more peripheral neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2021-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerin B Adelson, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (21):
- United States (21):
  - University of Connecticut, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Cleveland Clinic-Weston, Weston, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Saint Luke's, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 118 patients were enrolled from 17 institutions between May 2010 and October 2013
Pre-assignment Details: 118 postmenopausal women with ER-positive metastatic breast cancer resistant to aromatase inhibitors (AIs) were randomized to fulvestrant alone (Arm A) or in combination with bortezomib (Arm B). Two patients randomized to Arm B never received protocol therapy. Of 59 patients randomized to fulvestrant alone, Arm A, 27 crossed over to receive fulvestrant plus bortezomib (Arm C) at progression on fulvestrant alone.
Groups:
- Arm A: Fulvestrant Alone: Patients received fulvestrant IM on day 1 (days -14, 1, and 15 of course 1 only). Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may crossover to Arm C.
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
- Arm B: Fulvestrant + Bortezomib: Patients received fulvestrant IM as in Arm A and bortezomib IV on days 1, 8, and 15. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given IV
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
- Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib: Patients who crossed over from Arm A received fulvestrant IM on day 1 and bortezomib IV on days 1, 8, and 15. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given IV
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
Period: Randomized Phase
Arm/Group | Arm A: Fulvestrant Alone | Arm B: Fulvestrant + Bortezomib | Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib
Started | 59 | 59 | 0
Completed | 59 | 57 | 0
Not Completed | 0 | 2 | 0
Period: Crossover Phase
Arm/Group | Arm A: Fulvestrant Alone | Arm B: Fulvestrant + Bortezomib | Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib
Started | 0 | 0 | 27
Completed | 0 | 0 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Fulvestrant: Patients received fulvestrant IM on day 1 (days -14, 1, and 15 of course 1 only). Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may crossover to Arm C.
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Arm A: Fulvestrant | Arm B: Fulvestrant + Bortezomib | Total
Number analyzed (Participants) | 59 | 57 | 116
Age, Continuous [Median (Full Range); unit: years] | 57 [31 to 83] | 59 [31 to 80] | 57 [31 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 57 | 116
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 59 | 57 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS) at 12 Months
Description: The number of patients, treated with fulvestrant alone and fulvestrant plus bortezomib, who remained progression-free (Arms A vs. B). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Fulvestrant: Patients received fulvestrant IM on day 1 (days -14, 1, and 15 of course 1 only). Courses were repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may have crossed over into another treatment group (Arm C).
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
- Arm B: Fulvestrant + Bortezomib: Patients received fulvestrant as in arm A and bortezomib IV on days 1, 8, and 15. Courses were repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given IV
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Arm A: Fulvestrant | Arm B: Fulvestrant + Bortezomib
Number analyzed (Participants) | 59 | 57
Participants | 8 | 16

2. Primary Outcome: Number of Participants With Progression Free Survival (PFS) at 6 Months
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Fulvestrant | Arm B: Fulvestrant + Bortezomib
Number analyzed (Participants) | 59 | 57
Participants | 16 | 22

3. Secondary Outcome: Clinical Benefit Rate (CBR) of Adding Bortezomib to Fulvestrant in Arm C
Description: This outcome measure determined if the addition of bortezomib to fulvestrant improved the clinical benefit rate (defined as objective response plus stable disease for at least 24 weeks from day+1). Clinical Benefit Rate (CBR) is defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
Time Frame: Up to 24 weeks
Population: # of participants randomized to Arm A (Fulvestrant alone) who crossed over to fulvestrant plus bortezomib at progression (Arm C) and had clinical benefit.
Measure: Count of Participants; unit: Participants
Groups:
- Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib: Patients received fulvestrant IV on day 1 and bortezomib IM on days 1, 8, and 15. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib
Number analyzed (Participants) | 27
Participants | 5

4. Secondary Outcome: Number of Participants Who Survived Until Study End (up to 7 Years)
Description: Tabulation of the number of participants who survived from the date of first treatment until study end (up to 7 years).
Time Frame: From first treatment day until study end, assessed up to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Fulvestrant Alone | Arm B: Fulvestrant + Bortezomib
Number analyzed (Participants) | 59 | 57
Participants | 39 | 42

5. Secondary Outcome: Progression Free Survival at 24 Weeks (Arm C)
Time Frame: At 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib
Number analyzed (Participants) | 27
Participants | 5

6. Secondary Outcome: Frequency of Most Common Toxicities
Description: Most common toxicities in the fulvestrant arm alone (Arm A) and the fulvestrant/bortezomib combination arm (Arm B). Most common toxicities are defined as adverse events having occurred in >10% of the participants within either (or both) Arm A or Arm B.
Time Frame: Up to 7 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Fulvestrant | Arm B: Fulvestrant + Bortezomib
Number analyzed (Participants) | 59 | 57
percentage of participants
  Hemoglobin-Low | 41 | 61
  White Blood Cell-Low | 32 | 42
  Hyperglycemia/Glucose-High | 44 | 51
  Hypoglycemia/Glucose-Low | 5 | 12
  SGOT (AST-High) | 25 | 32
  SGPT (ALT-High) | 14 | 21
  Neutrophil Count Decreased/ANC-low | 10 | 12
  Platelet Count Decreased/Platelets-Low | 8 | 30
  Hypocalcemia/Calcium-Low | 10 | 12
  Hyponatremia/Sodium-Low | 8 | 12
  Nausea | 29 | 63
  Vomiting | 14 | 32
  Diarrhea | 8 | 47
  Constipation | 34 | 46
  Heartburn/Dyspepsia | 10 | 18
  Anorexia | 15 | 23
  Headache | 12 | 25
  Pain (general) | 59 | 54
  Peripheral Neuropathy (Motor, Pain, Sensory) | 31 | 49
  Injection Site Reaction | 24 | 12
  Dyspnea | 32 | 19
  Cough | 29 | 23
  Fatigue | 56 | 56
  Limb Edema | 19 | 37
  Insomnia | 25 | 35
  Hot Flashes | 37 | 32
  Dizziness | 7 | 19
  Arthralgia | 36 | 28
  Myalgia | 10 | 18
  Anxiety | 8 | 19
  Fever | 15 | 12
  Pruritis | 7 | 16
  Rash/Desquamation | 8 | 11
  Depression | 8 | 16
  Anemia | 32 | 42
  Dry Eye | 0 | 12
  Hypertension | 12 | 21
  Rash (General) | 7 | 23
  Eye Disorders (not otherwise specified) | 7 | 12
  Urinary Disorders (General) | 15 | 11
  Thrombocytopenia | 41 | 61
  Neutropenia | 8 | 30
  Upper Respiratory Disorders (General) | 12 | 23
  Musculoskeletal Pain Disorders (not otherwise specified) | 17 | 18
  Mucositis Oral | 8 | 11

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: A 5% frequency threshold was set for the reporting of non-Serious Adverse Events (NSAEs) for this study. If the occurrence of an adverse event was observed in >5% of participants in any of the three treatment arms the event was reported for all three arms.
Groups:
- Arm A: Fulvestrant Alone: Patients received fulvestrant IM on day 1 (days -14, 1, and 15 of course 1 only). Courses were repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease may have crossed over to another treatment group (Arm C).
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
- Arm B: Fulvestrant + Bortezomib: Patients received fulvestrant IM as in Arm A and bortezomib IV on days 1, 8, and 15. Courses were repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given IV
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
- Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib: Patients who crossed over from Arm A at progression received fulvestrant IM on day 1 and bortezomib IM on days 1, 8, and 15. Courses were repeated every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given IV
  Fulvestrant: Given IM
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Arm A: Fulvestrant Alone | Arm B: Fulvestrant + Bortezomib | Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib
All-Cause Mortality (participants affected / at risk) | 11/59 | 15/57 | 9/27
Serious Adverse Events (participants affected / at risk) | 9/59 | 6/57 | 5/27
Other Adverse Events (participants affected / at risk) | 59/59 | 57/57 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Fulvestrant Alone (N=59) | Arm B: Fulvestrant + Bortezomib (N=57) | Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib (N=27)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — CTCAE Grade 5, unrelated to study drug
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) — CTCAE Grade 3
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) — CTCAE Grade 3
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — CTCAE Grade 4
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — CTCAE Grade 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — CTCAE Grade 3
Cardiac Disorder (Unspecified) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — CTCAE Grade 3
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — CTCAE Grade 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) — CTCAE Grade 3
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — CTCAE Grade 3
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — CTCAE Grade 3
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — CTCAE Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Fulvestrant Alone (N=59) | Arm B: Fulvestrant + Bortezomib (N=57) | Arm C: Crossover From Arm A at Progression to Fulvestrant + Bortezomib (N=27)
Anxiety (Psychiatric disorders) | 5 | 11 | 4
Depression (Psychiatric disorders) | 5 | 9 | 5 — Verbatim Terms: Depression, Seasonal Depression
Anemia (Blood and lymphatic system disorders) | 19 | 24 | 12
Neutropenia (Blood and lymphatic system disorders) | 5 | 17 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 35 | 15
Hyperglycemia (Metabolism and nutrition disorders) | 25 | 29 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 7 | 2
SGOT_AST-High (Metabolism and nutrition disorders) | 15 | 18 | 6
SGPT_ALT-High (Metabolism and nutrition disorders) | 8 | 12 | 5
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6 | 2
Nausea (Gastrointestinal disorders) | 16 | 34 | 12
Vomiting (Gastrointestinal disorders) | 7 | 17 | 6
Diarrhea (Gastrointestinal disorders) | 5 | 27 | 14
Constipation (Gastrointestinal disorders) | 20 | 26 | 11
Heartburn/Dyspepsia (Gastrointestinal disorders) | 6 | 10 | 1
Anorexia (Gastrointestinal disorders) | 9 | 13 | 4
Headache (Nervous system disorders) | 7 | 14 | 7
Pain (Nervous system disorders) | 35 | 31 | 10
Peripheral Neuropathy (Nervous system disorders) | 18 | 28 | 8 — Verbatim Terms: Neuropathy-Pain; Neuropathy-Motor; Neuropathy-Sensory
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 5 | 6 | 3
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 14 | 7 | 4
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 9 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 11 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 16 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10 | 4
Fatigue (General disorders) | 33 | 32 | 11
Limb Edema (General disorders) | 11 | 21 | 7
Fever (General disorders) | 9 | 7 | 1
Insomnia (General disorders) | 15 | 20 | 6
Dizziness (General disorders) | 4 | 11 | 3
Hot Flashes (General disorders) | 22 | 18 | 6
Creatinine increased (Investigations) | 2 | 4 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 7 | 2
Neutrophil Count Decreased (Investigations) | 6 | 7 | 0 — Absolute Neutrophil Count - low (Verbatim Term)
Infection with unknown Absolute Neutrophil Count (Infections and infestations) | 5 | 4 | 1 — Verbatim Term
Chills (General disorders) | 4 | 4 | 0 — Verbatim Term - Rigors/chills
Creatinine-Low (Investigations) | 2 | 3 | 0 — Verbatim Term
Total Bilirubin Low (Investigations) | 3 | 1 | 1 — Verbatim Term
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Blurred Vision (Eye disorders) | 0 | 5 | 1 — Verbatim Terms: Blurred Vision, Vision Changes
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0 | 2 — Verbatim Terms: Chronic Kidney Disease, Chronic Renal Disease
Dry Eye (Eye disorders) | 0 | 7 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Dysgeusia (Nervous system disorders) | 0 | 3 | 1 — Verbatim Terms: Dysgeusia, Taste Changes
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0
Flu Like Symptoms (General disorders) | 2 | 3 | 0 — Verbatim Terms: Flu Like Symptoms, Flu Symptoms, Flu Like Feeling
Hypertension (Vascular disorders) | 7 | 12 | 8 — Verbatim Terms: Hypertension, Hypertension-transient, High Blood Pressure
Malaise (General disorders) | 1 | 4 | 1
Mucositis Oral (Gastrointestinal disorders) | 5 | 6 | 3 — Verbatim Terms: Mouth Sore, Mucositis Oral, Mucositis, Mucosal Infection (System Organ Class: Infections and Infestations)
Numbness - fingers (Nervous system disorders) | 4 | 0 | 0 — General finger/hand numbness due to either Reynaud's syndrome or carpal tunnel
Rash (General, not otherwise specified) (Skin and subcutaneous tissue disorders) | 4 | 13 | 3 — Verbatim Terms: Rash Acneiform, Rash Maculo-papular, Purpura, Perioral Swelling, Skin Hyperpigmentation, Skin Redness, Shingles, Papulopustular Rash (Infections and Infestations - System Organ Class)
Pressure - left pubic area (Renal and urinary disorders) | 0 | 4 | 0 — Verbatim Term
Weight Loss (Investigations) | 4 | 2 | 5
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 — Verbatim Terms: Laryngeal Inflammation, Sore Throat
Toothache (Gastrointestinal disorders) | 2 | 1 | 2
Eye Disorders (not otherwise specified) (Eye disorders) | 4 | 7 | 3 — Verbatim Terms: Stye(s), Eyelid Function Disorder, Sore on Eyelid/Pruritis, Watering Eyes, Excessive Tearing (Right Eye), Glaucoma, Periocular Swelling, Cellulitis (Right Eye), Eye Infection (System Organ Class: Infections and Infestations)
Urinary Disorders (General) (Renal and urinary disorders) | 9 | 6 | 2 — Verbatim Terms: Urinary Frequency, Urinary Incontinence, Urinary Retention, Urinary Tract Obstruction, Urinary Urgency, Urine Odor, Urinary Tract Infection (System Organ Class: Infections and Infestations)
Reproductive system and breast disorders (General) (Reproductive system and breast disorders) | 5 | 1 | 1 — Verbatim Terms: Vaginal Discharge, Vaginal Dryness, Vaginal Hemorrhage, Vaginal Odor, Vulval Infection (System Organ Class: Infections and Infestations), Vaginal Infection (System Organ Class: Infections and Infestations), Bacterial Vaginosis
Upper Respiratory Disorders (General) (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 8 — Verbatim: Allergic Rhinitis, Nasal Congestion, Sinus Disorder/Common Cold, Sinus Congestion, Rhinorrhea, Seasonal Allergies (sinus). Sinusitis, Respiratory Infection and Upper Respiratory Infection (System Organ Class: Infections and Infestations)
Lower Respiratory Disorders (General, not otherwise specified) (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 — Verbatim Terms: Pneumonitis, Asthma, Bronchospasm, Hemoptysis, Bronchial Infection (System Organ Class: Infections and Infestations), Pleural Infection (System Organ Class: Infections and Infestations)
Ear Disorders (General) (Ear and labyrinth disorders) | 2 | 1 | 2 — Verbatim Terms: Ear Pain, Ear Fullness/Pressure, Tinnitus, Otitis Media (System Organ Class: Infections and Infestations)
Skin Infections (General) (Infections and infestations) | 3 | 3 | 3 — Verbatim Terms: Skin Infection, Skin Infection (Viral), Skin Infection (insect bite), Cellulitis, Cellulitis around pleurex site
Infections (General), not otherwise specified (Infections and infestations) | 3 | 4 | 1 — Verbatim Terms: Infection, Infection localized (big toe), Infection (other), Lip Infection, Nail Infection, Soft Tissue Infection, Herpes
Musculoskeletal Pain Disorders (not otherwise specified) (Musculoskeletal and connective tissue disorders) | 10 | 10 | 7 — Verbatim: Generalized Muscle Weakness, Muscle Cramping, Muscle Spasms, Muscle Tension, Muscle Cramping - back, Muscle Weakness - lower limb, Pain - left deltoid muscle, Leg Cramps, Leg Pain, Bone Pain, Jaw Clicking, Osteonecrosis-Jaw, Neck Tightness
Sinus Tachycardia (Cardiac disorders) | 2 | 0 | 2 — Verbatim Terms: Sinus Tachycardia, Rapid Heartbeat
Carcinomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 — Verbatim Terms: Basal Cell Carcinoma, Squamous Cell Carcinoma
Hemoglobin - Low (Blood and lymphatic system disorders) | 24 | 35 | 15
White Blood Cells Decreased (Investigations) | 19 | 24 | 12
Platelet Count Decreased (Investigations) | 5 | 17 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less